CLINICAL TRIAL: NCT06350539
Title: Personalized Models for Cancer Research
Status: Recruiting | Type: Observational
Sponsor: New York Stem Cell Foundation Research Institute (Other)
Collaborators: Stevens Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 10-007
Record Dates: First submitted 2024-03-21; First posted 2024-04-05 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumor, Adult
Keywords: cancer; solid tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Affected Subjects: Subjects in this group will have a solid tumor cancer diagnosis.
  Interventions: Other: Biological Sample Collection
- Healthy Control: Subjects in this group will serve as healthy controls.
  Interventions: Other: Biological Sample Collection

INTERVENTIONS:
Other: Biological Sample Collection — Excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure).

SUMMARY:
The New York Stem Cell Foundation (NYSCF) Research Institute is performing this research to accelerate cancer research ranging from disease mechanisms to personalized medicine approaches that will help to realize the promise of precision medicine for oncology.

DETAILED DESCRIPTION:
Researchers at the New York Stem Cell Foundation (NYSCF) Research Institute will establish a living biobank of tumor/organoids and stem cells representing individual patients diagnosed with cancer. Samples from healthy individuals (non-cancer diagnosis) or from non-disease tissue will also be collected to be used as controls in this study.

Information and biospecimens may be transferred to NYSCF by external institution or NYSCF research personnel may prospectively enroll participants to have portions of samples or cells that were (or will be) collected for reasons other than this study transferred into the biobank.

NYSCF's researchers hypothesize that the development of patient-specific models that can expand in vitro while capturing tumor complexity at the genotypic and phenotypic levels will enable accelerated discovery of more efficient treatments for patients and improve outcomes.

This study is not a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 and older with a solid tumor cancer diagnosis.
* Adults ages 18 and older serving as healthy controls.

Exclusion Criteria:

* Human fetuses.
* Neonates.
* Children.
* Wards of the state.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a solid tumor cancer diagnosis or adults without a medical condition to serve as healthy controls (a comparison group for those with a solid tumor cancer diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2034-02-15 (Estimated); Study Completion 2034-02-15 (Estimated)

PRIMARY OUTCOMES:
Implement organoid culture technologies. | Baseline
  NYSCF will establish patient specific tumor models known as organoids. Organoids are three dimensional cell culture laboratory models with self-organizing capabilities and long-term expansion potential that recapitulate the tissue they are derived from at the histological, molecular, and phenotypic level. We will create organoids from each subject sample collected. Primary outcome measure is successful growth of organoids from individual tumor samples.
Validate genotypic and phenotypic relevance of tumor-derived organoids for biobanking. | Baseline
  To ensure the validity of outcome 1, NYSCF will perform a series of molecular and histological evaluations in primary tissues versus the derived organoid model.
Establish functional testing using organoid cultures alone or in combination with additional cell types. | Baseline
  To validate the clinical utility of the organoid models and the discovery of novel therapeutic strategies, NYSCF will establish methodologies to evaluate organoid responses (i.e., genetic, phenotypic, morphological changes) to small molecules and/or additional treatment modalities such as immunotherapies, antibody-based therapeutics, and others.
Perform drug testing and screens to identify new targets and/or new therapeutic strategies to effectively treat cancer. | Baseline
  As with outcome 3, to validate the clinical utility of the organoid models and the discovery of novel therapeutic strategies, NYSCF will establish methodologies to evaluate organoid responses (i.e., genetic, phenotypic, morphological changes) to small molecules and/or additional treatment modalities such as immunotherapies, antibody-based therapeutics, and others.
Develop a Laboratory Developed Test (LDT) for CLEP/FDA approval that will inform clinicians of each patient's tumor responses to FDA approved drugs. | Baseline
  Tumor organoid models have been shown to recapitulate patient's responses to certain chemotherapies, radiation, and combination regimens used as standard of care. These models hold an unprecedented potential to predict patient's responses preclinically and become an additional resource that clinicians can use to inform treatment decisions. NYSCF will adapt the methodology developed in Outcome 4 to an assay performed under clinical laboratory standards and regulation to pursue clinical certification/FDA approval as per regulatory requirements.
Develop stem cells from individual patient samples to study tumor evolution. | Baseline
  Induced pluripotent stem cells are an invaluable source of patient material with unlimited self-renewal potential that can be used to generate any cell type in the body. By creating iPSCs from each patient's material received at our labs, NYSCF will generate the relevant cell tissue type to study the contribution of germline genetic risk factors to the development of each patient's specific cancers so that we can understand the mechanisms driving tumor evolution and adaptation to therapies as well as the potential of environmental factors and/or the role of immune surveillance that may determine the development of malignant disease. These studies may also lead to the identification of biomarkers for early detection and/or for more effective surveillance before recurrence occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Andres-Martin, PhD, Principal Investigator — New York Stem Cell Foundation Research Institute
Locations (1):
- New York Stem Cell Foundation Research Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No